CLINICAL TRIAL: NCT02369588
Title: Effects of Portion Size of Multiple Items at a Meal on Food Intake of Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PortionSize102; R01DK059853 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Feeding Behaviors
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100% Portion Sizes (Experimental): Food portion size Test meal consists of baseline (100%) portion size of all foods
  Interventions: Other: Food portion size
- 133% Portion Sizes (Experimental): Food portion size Test meal consists of portion sizes of all foods that are 133% the size of baseline portions
  Interventions: Other: Food portion size
- 167% Portion Sizes (Experimental): Food portion size Test meal consists of portion sizes of all foods that are 167% the size of baseline portions
  Interventions: Other: Food portion size
- 200% Portion Sizes (Experimental): Food portion size Test meal consists of portion sizes of all foods that are 200% the size of baseline portions
  Interventions: Other: Food portion size

INTERVENTIONS:
Other: Food portion size

SUMMARY:
This study tests the effect of serving larger portions of all foods in a meal on the outcome of food and energy intake. Using a crossover design, participants are served the meal once a week for four weeks and the portion sizes are varied at each meal. Some of the foods served at the meal are low in calorie density (calories per gram) and some are higher in calorie density. The aim is to determine whether intake in response to larger portions differs depending on characteristics of the subjects or of the foods.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18 to 40 kg/square meter
* Regularly eat three meals per day
* Willing to eat foods served at test meals

Exclusion Criteria:

* Food allergies or restrictions
* Dieting to gain or lose weight
* Taking medications known to affect appetite
* Smoker
* Athlete in training
* Currently pregnant or breast-feeding
* Questionnaire score indicative of depression
* Questionnaire score indicative of disordered eating attitudes

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Differences in meal food intake | Weeks 1, 2, 3, and 4
  Differences in weight of food consumed (grams) at the meals
Differences in meal energy intake | Weeks 1, 2, 3, and 4
  Differences in energy of food consumed (kilocalories) at the meals
Differences in meal energy density | Weeks 1, 2, 3, and 4
  Differences in energy density of food consumed (kilocalories per gram) at the meal

SECONDARY OUTCOMES:
Differences in hunger and satiety | Weeks 1, 2, 3, and 4
  Differences in ratings of hunger and satiety either before or after the meal, as assessed by 100-mm visual analog scales (mm)
Differences in ratings of food properties | Weeks 1, 2, 3, and 4
  Differences in ratings of food properties (such as taste or healthfulness) as assessed either by 100-mm visual analog scales (mm) or ranking (rank order)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Rolls, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Roe LS, Kling SMR, Rolls BJ. What is eaten when all of the foods at a meal are served in large portions? Appetite. 2016 Apr 1;99:1-9. doi: 10.1016/j.appet.2016.01.001. Epub 2016 Jan 5. PMID 26767612